CLINICAL TRIAL: NCT03718819
Title: Effects of Combined Exercises on Postural Control With and Without Dual Task in Patients With Multiple Sclerosis
Brief Title: Effects of Exercises in MS on Postural Control With Dual Task
Acronym: MScombined
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Melda Soysal Tomruk, Principal investigator, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MST0047
Record Dates: First submitted 2018-10-16; First posted 2018-10-24 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; pilates; aquatherapy; postural control; dual task
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: exercise — Pilates and aquaplyometric exercises will be done combinedly.

SUMMARY:
Multiple sclerosis is a progressive neurological disease that associated with demyelinization and axonal damage. Decreased postural control is one of the initial symptom of disease. Improving postural control in people with neurological impairment is a common goal of physiotherapy. Doing exercises in water or land are examples for effective solutions. Pilates and aquaplyometric exercises are some of these approaches.

Performing daily activities at the same time requires dual tasking or multi tasking. Dual tasking is frequently impaired in MS. The aim of the study was to determine effect of combined Pilates and Aquaplyometric exercises on postural control with or without dual task in patients with multiple sclerosis.

DETAILED DESCRIPTION:
MS patients with decreased postural control will be enrolled eight-week, 45 minutes combined Pilates and aquaplyometric exercise programme. Postural control, hand dexterity and other functional parameteres will assess besaline and at the eighth week of exercise programme by the physiotherapist. Postural control will evaluate with and without dual task.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years old
* ability to walk independently or with single walking aid
* having stable symptoms

Exclusion Criteria:

* being acute or unstable phase of disease
* having EDSS score>6
* insuitable for the pool (incontinance, dermatological disease etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in limits of stability parameter with Biodex Balance System | Baseline and 8 weeks
  measured with Biodex Balance System (BBS; SD 12.1"Display 115 VAC). Patients were asked to stand on the rigid surface with barefoot and eyes open during measuring limits of stability. During each test trial, patients must shift their weight to move the cursor from the center target to a blinking target and back as quickly and with as little deviation as possible. The same process is repeated for each of the nine targets. Targets on the screen blink in random order. The tests repeated three times with 30 second resting time between trials. Patients' performance is evaluated from a total score of 100 where the higher score represents better trunk control.
Change in limits of stability parameter with cognitive task by Biodex Balance System | Baseline and 8 weeks
  Patients are asked to perform previously explained test protocol while maintaining balance they need to count down three-by-three from a randomly selected two-digit number. . Patients' performance is evaluated from a total score of 100 where the higher score represents better trunk control.

SECONDARY OUTCOMES:
Change in Nine hole peg Test | Baseline and 8 weeks
  The patient is seated at a table with a plastic NHPT placed at the patient's middle and asked to place pegs in a random order as quick as possible by using dominant hand first total time was recorded in seconds. Three consecutive trials with the dominant hand are immediately followed by three consecutive trials with the non-dominant hand.
Change in timed up and go test | Baseline and 8 weeks
  test was used to assess mobility and static and dynamic balance. The starting point was determined after the patient had been seated in a standart height chair with their back flush against the chair and their arms resting on the arm rests. The patients asked to stand up, walk three meters, turn around, walk back to the chair and sit down again. During the test the patients was expected to wear their regular footwear and use any mobility aids that they would normally require. Timing began when the patient started to rise and ended when returned to the chair and sit down. Lower time score represents better mobility and balance.
Change in 5-Repetititon Sit-To-Stand Test | Baseline and 8 weeks
  test is a meaure of the time taken to complete five repetitions of the STS movement. The patients were told to start the test in a seated position with full weight on the chair and arms folded across the chest. The feet were placed parallel to each other. The patients asked to move to a standing position with full knee extention and then back to a seated position as quickly as possible. After completion of five repetitions the test ended when patient touched the seat. Lower time score represents better lower extremity muscle strength
Change in timed 25 step walking test | Baseline and 8 weeks
  The patients were directed to one end of a clearly marked 25-foot course and was instructed to walk 25 feet as quickly as possible but safely. The time was calculated from the initiation of the instruction to start and ended when the patient had reached the 25-foot mark. Lower time score represents better walking or mobility performance
Handgrip strength test | Baseline and 8 weeks
  The patient was seated at a table and the subject holded the dynamometer in the dominant hand with the arm at right angles (90˚ flexion) and the elbow by the side of the body. The handle of the dynamometer was adjusted as the base should rest on first metacarpal, while the handle should rest on middle of four fingers. When ready the patient asked to squeeze the dynamometer with maximum isometric effort, which was maintained for about 5 seconds. Three consecutive trials were done and higher score was recorded (25). Higher score represents better grip force.

CONTACTS AND LOCATIONS:
Overall Officials: Barış Gürpınar, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, School of Physical Therapy and Rehabilitation, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
via clinical study
Supporting Information: CSR
Time Frame: in 2 years